CLINICAL TRIAL: NCT01200199
Title: Performance of Daily Electronic Diary to Capture Venous Symptoms Before and After Intervention for Great Saphenous Vein Incompetence
Brief Title: Validity of Electronic Diary for Monitoring Varicose Veins Symptoms
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: RS-002
Record Dates: First submitted 2010-09-08; First posted 2010-09-13 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Varicose veins

SUMMARY:
The purpose of this study is to contribute to the validation of an electronic daily diary to assess symptoms in patients with varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent and complete study assessments in written English
* Male or female age 18 to 75
* Patients having Saphenofemoral Junction (SFJ) incompetence and scheduled to receive foam sclerotherapy treatment for varicose veins in one leg
* Screening Symptom score of 7 points or more as measured by Question 1 on the modified VEINES-QOL/Sym questionnaire

Exclusion Criteria:

* Unable to comply with completing a daily diary for a total of 24 days
* Participation in any other investigational pharmaceutical product, or device study within the 3 months prior to Visit 1
* Current venous leg ulcer in either leg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Varicose veins
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility, variability, validity and sensitivity of patient's varicose vein symptoms using a disease-specific symptom questionnaire, administered as a daily electronic diary in patients undergoing treatment for varicose veins | 8 weeks

SECONDARY OUTCOMES:
To establish the treatment effect size of foam sclerotherapy treatment | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Wright, MD, Study Director — BTG International Inc.
Locations (1):
- Birmingham, United Kingdom